CLINICAL TRIAL: NCT03672929
Title: Allofit® IT With HXPE in Total Hip Arthroplasty. A Multi-center, Prospective, Non-controlled Post Market Surveillance Study
Brief Title: Allofit® IT With HXPE in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2010-25H
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Avascular Necrosis; Osteoarthritis, Hip; Inflammatory Arthritis; Post-Traumatic Osteoarthritis of Hip
Keywords: Total hip arthroplasty; Medical Device; Safety; Hip prosthesis
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the Allofit IT with HXPE: Subjects in need of a primary total hip arthroplasty, who met the inclusion/exclusion criteria and who received the Allofit IT Shell in combination with the Longevity HXPE Liners

SUMMARY:
The study design is a multi-center, prospective, non-controlled, consecutive cohort postmarket clinical follow-up study to obtain survival and outcome data on the Allofit IT Shell in combination with Longevity Liners in primary total hip arthroplasty.

DETAILED DESCRIPTION:
The study will involve orthopedic surgeons skilled in total hip arthroplasty and experienced with the implants subject of this study. In total, 5 centers will be involved. This number of clinical sites will permit assessment of the consistency among a multitude of Investigators. A total number of 200 subjects will be included in the study. It is anticipated that each clinical site will enroll 40-60 eligible study subjects, who have provided written informed consent.

Ethics Committee (EC) approval for each site has to be obtained prior to conducting this research. Sequentially, all eligible patients will be offered study enrollment at each center to avoid potential selection bias. All potential subjects will be required to participate in an informed consent process and sign an EC approved written informed consent prior to study enrollment. It is anticipated the enrollment period may be 12 months or longer to assure an adequate number of cases at each site. Each case enrolled will receive an Allofit IT HXPE Bearing System. The study is designed to be prospective to ensure that the study population is representative of the type of population that the device is intended to treat. The subjects included will be candidates for All subjects will undergo preoperative clinical, functional and radiographic evaluations, total hip arthroplasty, immediate post-operative evaluations and post-operative clinical, functional and radiographic evaluations at 6 months (± 1 month), 1 year (± 2 months), 2 year (± 2 months), 3 year (± 2 months), 5 year (± 2 months), 7 year (± 2 months), and 10 year (± 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN)
  * Osteoarthritis (OA)
  * Inflammatory arthritis (i.e. Rheumatoid arthritis)
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) of the affected hip joint(s).
* Patient has a Harris Hip Score <70 in the affected hip
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant.
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has a vascular (large and small vessel disease) insufficiency.
* The patient has a neurologic condition in the ipsalateral or contralateral limb which affects lower limb function.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give informed consent, or to comply with the follow-up program.
* The patient has received an investigational drug or device within the previous 6 months.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has osteoradionecrosis in the operative hip joint
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.
* The patient has known local bone tumors in the operative hip.
* The patient is Grade III obese with a Body Mass Index (BMI) > 40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of 200 males and females who require primary total hip arthroplasty. Subjects must be geographically accessible throughout the study and be willing and able to attend required follow-up appointments. Candidates who express interest in study participation will be offered informed consent, and eligibility will be determined based on the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2011-06-05 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (5):
- Medizinische Universität Wien, Universitätsklinik für Orhopädie, Vienna, Austria
- Service Clinique Chirurgicale Orthopédique et Traumatologique de l'hôpital "Hotel-Dieu", Nantes, France
- Germany (2):
  - Klinik Vincentium, Augsburg
  - Kliniken Dr. Erler, Nuremberg
- Traumatoloy and Orthopaedic Surgery, Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this study was initiated in 2011 and was completed in 2017. Medizinische Universitat Wien, Universitatsklinik fur Orthopadie, Austria enrolled 41 patients, CHU de Nantes - Site Nord, France enrolled 36 patients, Kliniken Dr. Erler GmbH, Germany enrolled 50 patients, Orthopadie El Masry, Germany enrolled 40 patients and HUA Santiago enrolled 30 patients
Pre-assignment Details: Enrollment for this study was initiated in 2011 and was completed in 2017 with 197 patients enrolled in five participating study centers. One site which enrolled 30 patients is inactive since a long time an only has data up to 1-year Post-OP.
Units Other Than Participants: implants
Period: Overall Study
Arm/Group | Patients Who Received the Allofit IT With HXPE
Started | 197; 197 implants
Completed | 98; 98 implants
Not Completed | 99; 99 implants
Not completed — Death | 13
Not completed — Lost to Follow-up | 32
Not completed — Withdrawal by Subject | 18
Not completed — Adverse Event | 3
Not completed — Surgery with the device never took place | 3
Not completed — Inactive site | 30

BASELINE CHARACTERISTICS:
Population: Demographic data were collected before surgery
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] — Age collected in years
  years | 63.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The gender for 2 participants is not available
  Participants
    number analyzed (Participants) | 195
    Female | 104
    Male | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 41
  France | 36
  Germany | 90
  Spain | 30
BMI [Mean (Standard Deviation); unit: kg/m²] — Body Mass Index Population: 1 patient does not have information on weight
  kg/m²
    number analyzed (Participants) | 196
    (all) | 28.0 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Survival of the Implant System
Description: The objective of this study is implant survival at 10 years which is assessed by revision of the the study device. Survivorship at 10 years was defined as cases that had the implant still in place at 10 years.
Time Frame: 10 years post-surgery
Population: All study patients
Measure: Number; unit: participants
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 197
participants | 89

2. Secondary Outcome: Safety of the Implant System
Description: Safety of the system will be assessed by monitoring the frequency and incidence of adverse events.
Time Frame: 10 years post-surgery
Population: 33 complications involved the study hip
Measure: Number; unit: complications
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 197
complications | 33

3. Secondary Outcome: Harris Hip Score (HHS)
Description: The Harris Hip Score (HHS) is an outcome measure that includes a series of questions answered by the patient and physical examinations recorded by a qualified health care professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). To obtain a final score, the points are summed. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: Due to lost to follow-up, withdrawals, visit not being performed the number of participants analyzed in each time-point is different
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 185
score on a scale
  Pre-Op | 51.5 (16.5)
  6 months: number analyzed (Participants) | 168
  6 months | 92.3 (10.0)
  1 Year: number analyzed (Participants) | 163
  1 Year | 94.4 (10.2)
  2 Year: number analyzed (Participants) | 122
  2 Year | 97.1 (6.0)
  3 Year: number analyzed (Participants) | 129
  3 Year | 96.6 (6.9)
  5 Year: number analyzed (Participants) | 103
  5 Year | 96.3 (8.1)
  7 Year: number analyzed (Participants) | 93
  7 Year | 93.0 (12.6)
  10 Year: number analyzed (Participants) | 86
  10 Year | 96.3 (7.8)

4. Secondary Outcome: EQ-5D-3L Score
Description: The EQ-5D-3L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes five dimensions referring to mobility, self-care, daily activities,pain/discomfort, and anxiety/depression. Each question can be answered in three ways/levels indicating no problems, some problems, and extreme problems. In the derived EQ-5D-3L score, the highest score is 1 and the lowest score is -0.594;negative numbers correspond to a self-assessed health state worse than being dead. Higher scores mean a better outcome.
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 193
score on a scale
  Pre-Op | 0.4 (0.3)
  6 months: number analyzed (Participants) | 173
  6 months | 0.9 (0.2)
  1 Year: number analyzed (Participants) | 164
  1 Year | 0.9 (0.2)
  2 Year: number analyzed (Participants) | 123
  2 Year | 0.9 (0.2)
  3 Year: number analyzed (Participants) | 132
  3 Year | 0.9 (0.2)
  5 Year: number analyzed (Participants) | 108
  5 Year | 0.9 (0.2)
  7 Year: number analyzed (Participants) | 96
  7 Year | 0.9 (0.2)
  10 Year: number analyzed (Participants) | 89
  10 Year | 0.9 (0.2)

5. Secondary Outcome: EQ-5D VAS
Description: The EQ-5D-3L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The VAS is a vertical scale ranging from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her current state of health. Higher scores mean a better outcome.
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 194
score on a scale
  Pre-Op | 52.7 (21.2)
  6 months: number analyzed (Participants) | 173
  6 months | 73.1 (19.7)
  1 Year: number analyzed (Participants) | 165
  1 Year | 78.4 (16.6)
  2 Year: number analyzed (Participants) | 121
  2 Year | 82.3 (13.6)
  3 Year: number analyzed (Participants) | 131
  3 Year | 82.1 (14.1)
  5 Year: number analyzed (Participants) | 109
  5 Year | 83.2 (16.3)
  7 Year: number analyzed (Participants) | 95
  7 Year | 81.9 (14.5)
  10 Year: number analyzed (Participants) | 88
  10 Year | 78.6 (16.8)

6. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27. Higher scores mean a better outcome.
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 194
score on a scale
  Pre-Op | 21.4 (7.4)
  6 months: number analyzed (Participants) | 174
  6 months | 41.1 (7.4)
  1 Year: number analyzed (Participants) | 167
  1 Year | 43.2 (6.4)
  2 Year: number analyzed (Participants) | 123
  2 Year | 44.8 (6.1)
  3 Year: number analyzed (Participants) | 132
  3 Year | 45.1 (5.4)
  5 Year: number analyzed (Participants) | 109
  5 Year | 45.5 (5.3)
  7 Year: number analyzed (Participants) | 96
  7 Year | 44.8 (6.7)
  10 Year: number analyzed (Participants) | 92
  10 Year | 45.5 (4.5)

7. Secondary Outcome: UCLA Activity Score
Description: The case administered University of California at Los Angeles (UCLA) score allows assessment of the case's activity level at each time point with scores from 1 (Wholly inactive: dependent on others; cannot leave residence) to 10 (Regularly participates in impact sports). Higher scores mean a better outcome
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 194
score on a scale
  Pre-Op | 4.3 (1.7)
  6 months: number analyzed (Participants) | 175
  6 months | 5.8 (1.8)
  1 Year: number analyzed (Participants) | 168
  1 Year | 6.0 (1.7)
  2 Year: number analyzed (Participants) | 124
  2 Year | 6.7 (1.3)
  3 Year: number analyzed (Participants) | 132
  3 Year | 6.7 (1.5)
  5 Year: number analyzed (Participants) | 109
  5 Year | 6.7 (1.7)
  7 Year: number analyzed (Participants) | 97
  7 Year | 6.6 (1.9)
  10 Year: number analyzed (Participants) | 93
  10 Year | 6.5 (1.8)

8. Secondary Outcome: Radiographic Evaluations - Acetabular Site
Description: X-rays evaluated for radiolucencies, osteolysis, hypertrophy, subsidence,heterotopic ossification, etc
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 196
Participants
  Immediat PostOp: Bone Condensation | 0
  Immediat PostOp: Cup migration | 1
  Immediat PostOp: Osteolysis | 0
  Immediat PostOp: Radiolucency | 6
  Immediat PostOp: None | 188
  Immediat PostOp: Screw breakage | 1
  6 Months: number analyzed (Participants) | 178
  6 Months: Bone Condensation | 0
  6 Months: Cup migration | 0
  6 Months: Osteolysis | 0
  6 Months: Radiolucency | 3
  6 Months: None | 175
  6 Months: Screw breakage | 0
  1 Year: number analyzed (Participants) | 174
  1 Year: Bone Condensation | 1
  1 Year: Cup migration | 1
  1 Year: Osteolysis | 0
  1 Year: Radiolucency | 1
  1 Year: None | 171
  1 Year: Screw breakage | 0
  2 Year: number analyzed (Participants) | 124
  2 Year: Bone Condensation | 1
  2 Year: Cup migration | 0
  2 Year: Osteolysis | 0
  2 Year: Radiolucency | 0
  2 Year: None | 123
  2 Year: Screw breakage | 0
  3 Year: number analyzed (Participants) | 133
  3 Year: Bone Condensation | 1
  3 Year: Cup migration | 0
  3 Year: Osteolysis | 0
  3 Year: Radiolucency | 1
  3 Year: None | 131
  3 Year: Screw breakage | 0
  5 Year: number analyzed (Participants) | 110
  5 Year: Bone Condensation | 1
  5 Year: Cup migration | 0
  5 Year: Osteolysis | 1
  5 Year: Radiolucency | 0
  5 Year: None | 108
  5 Year: Screw breakage | 0
  7 Year: number analyzed (Participants) | 96
  7 Year: Bone Condensation | 0
  7 Year: Cup migration | 0
  7 Year: Osteolysis | 0
  7 Year: Radiolucency | 0
  7 Year: None | 96
  7 Year: Screw breakage | 0
  10 Year: number analyzed (Participants) | 94
  10 Year: Bone Condensation | 0
  10 Year: Cup migration | 0
  10 Year: Osteolysis | 0
  10 Year: Radiolucency | 0
  10 Year: None | 94
  10 Year: Screw breakage | 0

9. Secondary Outcome: Radiographic Evaluations - Femoral Side
Description: X-rays evaluated for radiolucencies, osteolysis, hypertrophy, subsidence,heterotopic ossification, etc
Time Frame: pre-op, 6 Months, 1 Year, 2 Year, 3 Year, 5 Year, 7 Year, 10 Year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Received the Allofit IT With HXPE
Number analyzed (Participants) | 196
Participants
  Immediat PostOp: Stem Shift | 0
  Immediat PostOp: Stem Subsidence Subsidence | 6
  Immediat PostOp: Calcar rounding | 5
  Immediat PostOp: Calcar resorption | 3
  Immediat PostOp: Abnormalities | 0
  Immediat PostOp: Heterotopic Ossification | 0
  Immediat PostOp: AP- View: Radiolucency | 1
  Immediat PostOp: AP- View: Osteolysis | 0
  Immediat PostOp: Lateral - View: Radiolucency | 0
  Immediat PostOp: Lateral - View: Osteolysis | 1
  Immediat PostOp: None | 180
  6 Months: number analyzed (Participants) | 179
  6 Months: Stem Shift | 1
  6 Months: Stem Subsidence Subsidence | 6
  6 Months: Calcar rounding | 55
  6 Months: Calcar resorption | 5
  6 Months: Abnormalities | 1
  6 Months: Heterotopic Ossification | 3
  6 Months: AP- View: Radiolucency | 2
  6 Months: AP- View: Osteolysis | 2
  6 Months: Lateral - View: Radiolucency | 0
  6 Months: Lateral - View: Osteolysis | 1
  6 Months: None | 103
  1 Year: number analyzed (Participants) | 174
  1 Year: Stem Shift | 3
  1 Year: Stem Subsidence Subsidence | 4
  1 Year: Calcar rounding | 68
  1 Year: Calcar resorption | 5
  1 Year: Abnormalities | 0
  1 Year: Heterotopic Ossification | 2
  1 Year: AP- View: Radiolucency | 6
  1 Year: AP- View: Osteolysis | 1
  1 Year: Lateral - View: Radiolucency | 0
  1 Year: Lateral - View: Osteolysis | 2
  1 Year: None | 83
  2 Year: number analyzed (Participants) | 124
  2 Year: Stem Shift | 1
  2 Year: Stem Subsidence Subsidence | 0
  2 Year: Calcar rounding | 62
  2 Year: Calcar resorption | 2
  2 Year: Abnormalities | 0
  2 Year: Heterotopic Ossification | 1
  2 Year: AP- View: Radiolucency | 5
  2 Year: AP- View: Osteolysis | 0
  2 Year: Lateral - View: Radiolucency | 1
  2 Year: Lateral - View: Osteolysis | 0
  2 Year: None | 52
  3 Year: number analyzed (Participants) | 133
  3 Year: Stem Shift | 1
  3 Year: Stem Subsidence Subsidence | 0
  3 Year: Calcar rounding | 56
  3 Year: Calcar resorption | 1
  3 Year: Abnormalities | 0
  3 Year: Heterotopic Ossification | 4
  3 Year: AP- View: Radiolucency | 5
  3 Year: AP- View: Osteolysis | 1
  3 Year: Lateral - View: Radiolucency | 3
  3 Year: Lateral - View: Osteolysis | 1
  3 Year: None | 61
  5 Year: number analyzed (Participants) | 110
  5 Year: Stem Shift | 1
  5 Year: Stem Subsidence Subsidence | 0
  5 Year: Calcar rounding | 50
  5 Year: Calcar resorption | 3
  5 Year: Abnormalities | 0
  5 Year: Heterotopic Ossification | 4
  5 Year: AP- View: Radiolucency | 6
  5 Year: AP- View: Osteolysis | 1
  5 Year: Lateral - View: Radiolucency | 1
  5 Year: Lateral - View: Osteolysis | 1
  5 Year: None | 43
  7 Year: number analyzed (Participants) | 96
  7 Year: Stem Shift | 0
  7 Year: Stem Subsidence Subsidence | 0
  7 Year: Calcar rounding | 52
  7 Year: Calcar resorption | 1
  7 Year: Abnormalities | 1
  7 Year: Heterotopic Ossification | 5
  7 Year: AP- View: Radiolucency | 6
  7 Year: AP- View: Osteolysis | 1
  7 Year: Lateral - View: Radiolucency | 0
  7 Year: Lateral - View: Osteolysis | 0
  7 Year: None | 30
  10 Year: number analyzed (Participants) | 94
  10 Year: Stem Shift | 0
  10 Year: Stem Subsidence Subsidence | 0
  10 Year: Calcar rounding | 45
  10 Year: Calcar resorption | 2
  10 Year: Abnormalities | 0
  10 Year: Heterotopic Ossification | 3
  10 Year: AP- View: Radiolucency | 5
  10 Year: AP- View: Osteolysis | 2
  10 Year: Lateral - View: Radiolucency | 1
  10 Year: Lateral - View: Osteolysis | 2
  10 Year: None | 34

ADVERSE EVENTS:
Time Frame: 10 years post-surgery
Description: Same definitions
Arm/Group | Patients Who Received the Allofit IT With HXPE
All-Cause Mortality (participants affected / at risk) | 13/197
Serious Adverse Events (participants affected / at risk) | 52/197
Other Adverse Events (participants affected / at risk) | 25/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Allofit IT With HXPE (N=197)
General (Cardiac disorders) | 8 (13) — Cardiovascular
General (Renal and urinary disorders) | 1 (1)
General (Infections and infestations) | 1 (1) — Infection non hip
General (Musculoskeletal and connective tissue disorders) | 17 (18) — muscoskeletal non hip
General (Nervous system disorders) | 1 (2)
General (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) — Oncological
General (Respiratory, thoracic and mediastinal disorders) | 2 (3) — Pulmonary
General (General disorders) | 10 (13)
Hip Related (Product Issues) | 2 (4) — Fracture of femur
Hip Related (Product Issues) | 3 (5) — Other Hip Related Radiographic Finding
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received the Allofit IT With HXPE (N=197)
General Complications - Adverse Events (Gastrointestinal disorders) | 2 (4)
General Complications - Adverse Events (Musculoskeletal and connective tissue disorders) | 8 (17) — muscuskeletal non hip
General Complications - Adverse Events (General disorders) | 3 (13) — other general complication
Hip Related Complications - Adverse Events (Product Issues) | 4 (8) — Dislocation
Hip Related Complications - Adverse Events (Vascular disorders) | 3 (3) — Hematoma
Hip Related Complications - Adverse Events (General disorders) | 2 (2) — Subluxation
Hip Related Complications - Adverse Events (General disorders) | 3 (3) — Pain

LIMITATIONS AND CAVEATS:
Over the pandemic many patients did not complete their visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-02-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03672929/Prot_SAP_ICF_000.pdf